CLINICAL TRIAL: NCT00938366
Title: An Open-label, Cross Over Study, to Assess the Interactions of Pantoprazole (Proton Pump Inhibitor) With Oral Cladribine Administered in Subjects With Multiple Sclerosis
Brief Title: Drug-Drug Interaction of Cladribine and Pantoprazole in Multiple Sclerosis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A., Geneva (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 27967
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cladribine followed by Cladribine + Pantoprazole (Experimental): Subjects will receive a single dose of cladribine10 milligram (mg) orally on Day 1. After a wash out period of 10-25 days, subjects will receive pantoprazole 40 mg orally for 2 consecutive days. On Day 2 of the pantoprazole administration, a single dose of cladribine 10 mg will be administered orally 3 hours after the second pantoprazole dose.
  Interventions: Drug: Cladribine; Drug: Pantoprazole
- Cladribine + pantoprazole followed by Cladribine (Experimental): Subjects will receive pantoprazole 40 mg orally for 2 consecutive days. On Day 2 of the pantoprazole administration, a single dose of cladribine 10 mg will be administered orally 3 hours after the second pantoprazole dose. After a wash out period of 10-25 days, subjects will receive a single dose of cladribine 10 mg orally.
  Interventions: Drug: Cladribine; Drug: Pantoprazole

INTERVENTIONS:
Drug: Cladribine — Subjects will receive two single doses of 10 mg cladribine orally in either first or second intervention period followed by a washout period of 10-25 days.
Drug: Pantoprazole — Subjects will receive a pantoprazole 40 mg orally for 2 consecutive days either in first or second intervention period.

SUMMARY:
The purpose of the study is to assess the influence of pantoprazole on the pharmacokinetic profile of cladribine, especially in terms of extent of absorption of cladribine since pH-modifying drug may potentially affect the stability of cladribine and thereby its bioavailability

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a body mass index less than or equal to (<=) 28 and have a body weight greater than (>) 60 kilogram (kg) and less than (<) 120 kg, at screening
* Able to understand informed consent and had given written, informed consent
* Had a diagnosis of clinically stable and definite multiple sclerosis (MS) by either McDonald or Poser criteria
* Expanded disability status scale (EDSS) score not to exceed 5.0
* Male or non-pregnant, non-breast feeding women aged 18 to 65 years, inclusive at the time that informed consent was obtained
* Female subjects lacking childbearing potential defined as post-menopausal for at least two years, surgically or medically sterile or sexually inactive; or willing to avoid pregnancy by using an adequate method of birth control for 28 days prior to, during and up to 90 days after the last administration of trial medication

Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Subjects presenting a severe or unstable disorder: poorly controlled diabetes or arterial hypertension, severe cardiac insufficiency, unstable ischemic heart disease, a significant pre-existing hematological disease, or any medical condition, which in the opinion of the investigator, would constitute a risk or a contraindication for the participation of the subject to the study or that could interfere with the study objectives, conduct or evaluation
* Subjects who were on MS treatment; and subjects who were on a non-stable symptomatic MS treatment (stable dose was defined as 3 weeks or longer prior to first study dose)
* Clinically significant abnormal laboratory test results or electrocardiogram findings that in the opinion of the investigator could increase the safety risk to the subject
* Positive results from serology examination for Hepatitis B surface antigen (HbsAg) not due to vaccination, hepatitis B core antibody (HbcAb), Hepatitis C virus antibody (anti-HCV) or Human Immunodeficiency antibody (anti-HIV)
* Signs and symptoms of Transmissible Spongiform Encephalopathy at screening, or family members who suffered from such
* Presence of chronic or recurrent infection or any acute infection within the last 2 weeks before first dosing in each study period
* Presence of gastrointestinal disease that, in the opinion of the investigator, could affect the pharmacokinetic outcome of the study
* Consumption of any concomitant medication that could directly influence gastric acidity (example: use of antacids, histamine receptor (H2) antagonists or other proton pump inhibitor) taken within 7 days of study day 1 and throughout the study period
* Intake of alcoholic beverages, caffeine and caffeine containing beverages, grapefruit, oranges, cranberries and juices of these three fruits or smoking in the 48 hours prior to first dose and 48 hours post dose (cladribine)
* Exposure to any investigational drug or the use of any investigational device in the 12 weeks prior to first dose
* Intake of any medications that could directly influence gastrointestinal motility and absorption of cladribine (example, use of H2-antagonists, proton pump inhibitors) 7 days prior to cladribine administration
* Any immunomodulatory therapy (including but not limited to glatiramer acetate, interferons, or natalizumab) and treatment with oral or systemic corticosteroids or adrenocorticotropic hormone within 28 days of first dosing
* Any cytokine or anti-cytokine therapy, IV immunoglobulin administration or plasmapheresis was prohibited in the 3 months prior to first dosing
* Current history or presence of drug or alcohol abuse, confirmed by positive test results for drugs of abuse and/or alcohol or had a history of drug or alcohol abuse. Alcohol abuse was defined as: an average daily intake of more than 3 units or a weekly intake of more than 21 for males and 14 units for females where 1 unit equals 8-10 gram alcohol (1 unit equals 340 milliliter [mL] of beer, 115 mL of wine or 43 mL of spirits)
* History or presence of hypertension or other significant cardiovascular abnormality, history of heart or kidney disease
* Current diagnosis or personal history of cancer
* Smoke 10 cigarettes or more per day or equivalent
* Loss or donation of more than 400 mL of blood in the 12 weeks prior to first dose.
* Definite or suspected personal history or family history of adverse drug reaction or hypersensitivity to drugs with a similar chemical structure to cladribine or pantoprazole or with known hypersensitivity to cladribine or pantoprazole excipients
* Presence or history of any serious allergy (requiring hospitalization or prolonged systemic treatment)
* Pregnant or nursing women. Treatment of pregnant and nursing women with cladribine in this study was prohibited
* Signs or symptoms of neurological disease other than MS that could explain the symptoms of the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, PhD, Study Director — Merck Serono S.A. - Geneva, an affiliate of MerckKGaA, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover study.18 subjects were included and washout of 10 to 25 days separated each treatment period. Overall 17 subjects completed the trial.1 subject withdrew consent after completion of the first period (cladribine alone) and was excluded from Pharmacokinetic population.18 subjects were included in safety population.
Groups:
- Cladribine Followed by Cladribine + Pantoprazole: Subjects received a single 10 milligram (mg) cladribine dose orally on Day 1 followed by a wash out period of 10-25 days. Subjects then received pantoprazole 40 mg orally for 2 consecutive days. A single 10 mg cladribine dose was administered orally after 3 hours of fasting post pantoprazole dose on second day. After administration of cladribine, subjects were required to fast for an additional 2 hours.
- Cladribine + Pantoprazole Followed by Cladribine: Subjects received pantoprazole 40 mg orally for 2 consecutive days. A single 10 mg cladribine dose was administered orally after 3 hours of fasting post the pantoprazole dose on second day. After a wash out period of 10-25 days, subjects received a single 10 mg cladribine dose orally.
Period: Overall Study
Arm/Group | Cladribine Followed by Cladribine + Pantoprazole | Cladribine + Pantoprazole Followed by Cladribine
Started | 9 | 9
Completed | 8 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized subjects.
Groups:
- Cladribine Followed by Cladribine + Pantoprazole: Subjects received a single 10 milligram (mg) cladribine dose orally on Day 1 followed by a wash out period of 10-25 days. Subjects then received pantoprazole 40 mg orally for 2 consecutive days. A single 10 mg cladribine dose was administered orally after 3 hours of fasting post the pantoprazole dose on second day. After administration of cladribine, subjects were required to fast for an additional 2 hours.
- Total: Total of all reporting groups
Arm/Group | Cladribine Followed by Cladribine + Pantoprazole | Cladribine + Pantoprazole Followed by Cladribine | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.56 (11.75) | 46.89 (8.31) | 45.72 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Cladribine
Description: The maximum or peak plasma concentration observed after the administration of cladribine.
Time Frame: Pre-dose (within 30 minutes prior to dosing) and at 0.5,1, 3, 6, 8, 12,16, 24, 36, 48 Hour post-dose
Population: Pharmacokinetic (PK) analysis set included all the subjects who received cladribine alone and cladribine + pantoprazole according to the randomization and completed the full PK sampling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Groups:
- Cladribine: Subjects received two single doses of cladribine 10 mg orally in either first or second intervention period followed by a washout period of 10-25 days.
- Cladribine + Pantoprazole: Subjects received pantoprazole 40 mg orally for 2 consecutive days. A single 10 mg cladribine dose was administered orally after 3 hours of fasting post the pantoprazole dose on second day in either first or second intervention period.
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 17 | 17
nanogram/milliliter | 20.7 (28.2) | 20.3 (46.0)

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Cladribine
Description: The AUC (0-t) was defined as the area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t).
Time Frame: Pre-dose (within 30 minutes prior to dosing) and at 0.5,1, 3, 6, 8, 12,16, 24, 36, 48 Hour post-dose
Population: The PK analysis set included all the subjects who received cladribine alone and cladribine + pantoprazole according to the randomization and completed the full PK sampling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 17 | 17
hour*nanogram/milliliter | 71.5 (28.0) | 71.3 (36.6)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Cladribine
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: Pre-dose (within 30 minutes prior to dosing) and at 0.5,1, 3, 6, 8, 12,16, 24, 36, 48 Hour post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 17 | 17
hour*nanogram/milliliter | 74.6 (27.7) | 75.0 (34.8)

4. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Cladribine
Description: The tmax was defined as time taken by the drug cladribine to reach Cmax.
Time Frame: Pre-dose (within 30 minutes prior to dosing) and at 0.5,1, 3, 6, 8, 12,16, 24, 36, 48 Hour post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 17 | 17
hour | 0.5 [0.5 to 1.0] | 0.6 [0.5 to 1.0]

5. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Cladribine
Description: The apparent terminal half-life was defined as the time required for the plasma concentration of drug cladribine to decrease 50 percent (%) in the final stage of its elimination.
Time Frame: Pre-dose (within 30 minutes prior to dosing) and at 0.5,1, 3, 6, 8, 12,16, 24, 36, 48 Hour post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 17 | 17
hour | 14.0 (18.2) | 14.9 (23.8)

6. Secondary Outcome: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of Cladribine
Description: Clearance of a drug was a measure of the rate at which cladribine is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose was influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose (within 30 minutes prior to dosing) and at 0.5,1, 3, 6, 8, 12,16, 24, 36, 48 Hour post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 17 | 17
liter/hour | 134.0 (27.7) | 133.3 (34.8)

7. Other Pre Specified Outcome: Apparent Volume of Distribution During the Terminal Phase Following Extravascular Administration (Vz/f) of Cladribine
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Pre-dose (within 30 minutes prior to dosing) and at 0.5,1, 3, 6, 8, 12,16, 24, 36, 48 Hour post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 17 | 17
liter | 2709 (32) | 2875 (46)

8. Secondary Outcome: Percentage of Subjects With Any Treatment Emergent Adverse Events (TEAEs), Serious AEs, AEs Leading to Death, and AEs Leading to Discontinuation
Description: An AE was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 1 year, that were absent before treatment or that worsened relative to pre treatment state. AEs Leading to Death and AEs Leading to Discontinuation were also presented in the outcome measure.
Time Frame: Up to 1 year
Population: Safety analysis set included all the randomized subjects who received treatment with at least one dose of either cladribine or pantoprazole during the study period.
Measure: Number; unit: percentage of subjects
Arm/Group | Cladribine | Cladribine + Pantoprazole
Number analyzed (Participants) | 18 | 17
percentage of subjects
  TEAEs | 11.1 | 0.0
  SAEs | 0.0 | 0.0
  AEs Leading to Death | 0.0 | 0.0
  AEs Leading to Discontinuation | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Cladribine | Cladribine + Pantoprazole
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 2/18 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine (N=18) | Cladribine + Pantoprazole (N=17)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other